CLINICAL TRIAL: NCT06876090
Title: Sarcopenia in Gestational Diabetes: The SiGnal-D Study
Brief Title: Sarcopenia in Gestational Diabetes
Acronym: SiGnal-D
Status: Recruiting | Type: Observational
Sponsor: Istituto di Neuroscienze Consiglio Nazionale delle Ricerche (Network)
Collaborators: University of Pisa (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andrea Tura, Principal Investigator, Istituto di Neuroscienze Consiglio Nazionale delle Ricerche
Other Study IDs: 2022XYXRJN_LS4_PRIN2022; B53D23022000006 (Other Grant/Funding Number: Italian Ministry of University and Research (in the context of Next Generation EU, Mission 4, Component 2))
Record Dates: First submitted 2025-03-03; First posted 2025-03-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia; Gestational Diabetes Mellitus (GDM); Pregnancy Complications; Adverse Maternal and Neonatal Outcomes; Cognitive Function
MeSH Terms: conditions — Sarcopenia; Diabetes, Gestational; Pregnancy Complications | interventions — Glucose Tolerance Test; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes (GDM) women
  Interventions: Diagnostic Test: Sarcopenia tests (for muscle mass, muscle function, physical performance); Diagnostic Test: Oral Glucose Tolerance Test; Other: Montreal Cognitive Assessment
- Pregnant women without gestational diabetes (non-GDM)
  Interventions: Diagnostic Test: Sarcopenia tests (for muscle mass, muscle function, physical performance); Diagnostic Test: Oral Glucose Tolerance Test; Other: Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Sarcopenia tests (for muscle mass, muscle function, physical performance) — We are not aware of any other study performing sarcopenia tests in GDM (or in pregnancy in general), with the aim of assessing sarcopenia prevalence in GDM/pregnancy, and related possible adverse pregnancy outcomes.
Diagnostic Test: Oral Glucose Tolerance Test — The OGTT, in combination with the sarcopenia tests, will allow to explore the relationships between the glucometabolic condition and the muscle quality in the pregnant women, either with GDM or with normal glucose tolerance.
Other: Montreal Cognitive Assessment — The MoCA questionnaire, in combination with the sarcopenia tests, will allow to explore the relationships between the cognitive function the presence of the sarcopenia syndrome in the pregnant women, either with GDM or with normal glucose tolerance.

SUMMARY:
Sarcopenia is a syndrome characterized by loss of skeletal muscle mass and strength, and physical performance deterioration. Prevalence of sarcopenia in elderly people is remarkably high (prevalence of about 25% in 60+ years people). In type 2 diabetes (T2D), sarcopenia is emerging as comorbidity of major concern. Sarcopenia, however, is not limited to elderly people, as it can develop also in younger individuals with prevalence around 9% or even higher according to some investigators. Of note, sarcopenia has been reported even in the 20-29 years interval. This interval includes women of childbearing age, thus raising the question whether sarcopenia may occur also in women with gestational diabetes (GDM) and whether this may affect pregnancy outcomes. Also, association between sarcopenia and cognitive impairment has been repeatedly reported, to the point that some authors have emphasized the importance of early sarcopenia recognition for prevention of cognitive impairment. Therefore, our main aims are:

1. To ascertain whether sarcopenia is present in GDM and, in that case, its prevalence;
2. To identify risk factors for sarcopenia;
3. To determine sarcopenia impact on pregnancy outcomes, and cognitive function.

During pregnancy, all women will undergo oral glucose tolerance test (OGTT) for assessment of the glucometabolic condition. Several clinical variables of interest in sarcopenia will also be recorded. As regards the OGTT data, special focus will be on the assessment of insulin resistance, both at fasting and during the dynamic conditions determined by the OGTT. Notably, the special interest for insulin resistance is due to the reason that this type of metabolic alteration is known to be a risk factor for sarcopenia. In fact, all women will then undergo testing for diagnosis of sarcopenia (or presarcopenia), and all data and parameters will be analyzed to identify relationships between sarcopenia-related variables and GDM-related ones. It is worth noting that in consideration of the exacerbated insulin resistance condition often observed in GDM, the investigators expect indeed a not negligible prevalence of sarcopenia (or at least presarcopenia) in GDM women, despite the young (non-elderly) age. In addition, since insulin resistance is often present in pregnancy even in the absence of dysglycemia, the investigators do not exclude to identify some cases of sarcopenia/presarcopenia even in pregnant non-GDM women. This study will be the basis for future studies (also of interventional type), especially in women with GDM for prevention of sarcopenia and related possible pregnancy complication and adverse pregnancy outcomes, as well as for possibly contributing to mitigation of risk for T2D development in later life.

ELIGIBILITY:
Inclusion Criteria:

At least one among the following conditions:

* Age equal to or higher than 35 years;
* Body mass index (BMI) equal to or higher than 25 kg/m^2;
* Glycemia between 5.6 and 6.9 mmol/L before or at the beginning of pregnancy;
* Fetal macrosomia in previous pregnancy;
* GDM in previous pregnancy;
* First-degree family history of diabetes.

Exclusion Criteria:

* Unmatching of at least one among the inclusion criteria;
* Twin pregnancy;
* Presence of any already known disease/disorder possibly affecting muscle mass or function;
* Neurological or psychiatric diseases;
* Already known diabetes (e.g., type 1 or type 2 diabetes).

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, based on the inclusion and exclusion criteria as outlined above.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sarcopenia/presarcopenia in pregnant women with and without gestational diabetes | Between week 28 and week 32 of pregnancy

OTHER OUTCOMES:
Identification of pre-gestational factors (obstetric history, pre-pregnancy body weight, dietary and physical activity habits) and gestational factors (body mass index, blood pressure, OGTT values) with risk of sarcopenia | Between week 16 and week 32 of pregnancy
  Pre-gestational data as well as gestational data, as indicated above, will be collected at visit V1 (week 16-18 for women at high GDM risk or week 24-28 for women not at high GDM risk), whereas sarcopenia diagnosis (visit V2) will occur between week 28 and 32 (sarcopenia diagnosis being necessary to indentify, among the indicated pre-gestational and gestational factors, the risk factors for sarcopenia itself).
Assessment of the potential impact of sarcopenia/presarcopenia on pregnancy outcomes (large or small for gestational age, LGA or SGA) | Between week 28 and week 32 of pregnancy
Exploration of the potential relationship between sarcopenia (presence or no presence of sarcopenia) and cognitive function in pregnancy (MoCA questionnaire score) | Between week 28 and week 32 of pregnancy
  The investigators will assess whether the MoCA questionnaire score is different in women with and without sarcopenia.
Assessment of the potential impact of sarcopenia/presarcopenia on pregnancy outcomes (type of delivery) | At the time of delivery

CONTACTS AND LOCATIONS:
Locations (3):
- Department of Obstetrics and Gynaecology, Division of Obstetrics and Feto-Maternal Medicine, Medical University of Vienna, Vienna, Vienna, Austria
- Italy (2):
  - Institute of Neuroscience, National Research Council, Padua, PD
  - Department of Clinical and Experimental Medicine, University of Pisa, Pisa, PI

IPD SHARING:
Plan to Share IPD: Undecided